CLINICAL TRIAL: NCT04416490
Title: A Prospective Observational Study to Investigate Patients' Prognosis and Patterns of Adjuvant Chemotherapy Use After Curative Resection of Primary Colon Cancer at High-risk Stage II or Stage III
Brief Title: Oxaliplatin Adjuvant Chemotherapy After Curative Resection of Primary Colon Cancer
Acronym: OCEAN
Status: Active, not recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-OXP-OS-401
Record Dates: First submitted 2020-04-27; First posted 2020-06-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stage II Colon Cancer; Stage III Colon Cancer
Keywords: colon cancer; high-risk stage; curative resection; adjuvant chemotherapy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with high-risk stage II or stage III primary colon cancer who have received curative resection

SUMMARY:
According to general medical guidelines, adjuvant chemotherapy is used after curative resection of high-risk stage II or III primary colon cancer. However, there exist limitations using clinical trial data acquired from highly selected subjects in a controlled environment. For example, patients aged over 70 years old were in many cases excluded from clinical trials resulting in insufficient data on the efficacy of therapies including oxaliplatin in aged patients, and the source data of the medical guidelines did not fully reflect the conditions of Korean patients. In addition, suggestions are continuously being submitted for existing therapies with modified administration periods and methods with the aim to search for the optimum effect over side effects. Discussions are also held on meta analyses results that imply the need to apply slightly different approaches through small groups of patient and disease factors. As there are more diverse adjuvant therapy protocols that can be applied to post-surgery colon cancer patients, it is necessary to figure out the patterns of adjuvant chemotherapies actually used in Korean medical practices. Also, in order to complement the limitation of external validity of the existing base clinical data, a multifaceted exploratory analysis will be conducted by making follow-up observations on patterns, prognosis results, quality of life, adverse effects, etc. of post-surgery adjuvant chemotherapies actually used in around 30 sites in Korea under the noninterventional observational study conditions.

DETAILED DESCRIPTION:
[Overview] Investigators will obtain voluntary consent for participation in this study from patients with high-risk stage II or stage III colon cancer who require or are planning to receive adjuvant chemotherapy after curative resection. Patients who provided written consent for using their personal information and who satisfy inclusion/exclusion criteria will be given a study enrollment number. Among the predefined study-relevant data, available data on these patients will be collected in the case report forms (CRF) until the study is completed.

[Follow-up observation schedule and the scope of data collection] Since this study is an observational study, data collection in the CRF will be restricted to the data created only from usual treatment practices and there will be no separate test or additional drug administration for the study. However, subjects will be asked to complete questionnaire to evaluate their quality of life at the following time points: baseline, Month 3 (13 weeks ± 2 weeks), Month 6 (26 weeks ± 2 weeks), Month 12 (52 weeks ± 4 weeks), Month 24 (104 weeks ± 8 weeks), Month 36 (156 weeks ± 8 weeks). For subjects who drop out from the study or in case of disease event (relapse, metastasis or new primary malignant tumor), the questionnaire will be conducted at the time of drop-out or disease event. Survival of all subjects (including those who drop out from the study or whose disease event is confirmed) will be checked every 6 months after adjuvant chemotherapy started. Among the data created from the subjects on their visits for treatment, the following data will be collected for the purpose of this study.

* Demographics of the subjects.
* Colon cancer information (diagnosis information, risk factors, surgery information).
* Whether or not neoadjuvant chemotherapy was conducted.
* Underlying disease.
* Adjuvant chemotherapy information.
* Other concomitant medication (drugs administered for prevention and treatment of OXLIPN, drugs administered for treatment of Grade 3-4 adverse drug reactions/serious adverse drug reactions related to the chemotherapy).
* Vital signs, height, and weight.
* Performance Status evaluation (ECOG PS).
* Geriatric Assessment (KG-7): for subjects ≥ 65 years old.
* Quality of Life assessment (FACT-C, FACT/GOG-NTX-12).
* Laboratory test results.
* Tumor Marker (CEA, CA 19-9) test results.
* Molecular genetic test results (MSI [microsatellite instability] and/or MMR [DNA mismatch repair gene], immunohistochemistry test for protein, KRAS, NRAS, BRAF etc.).
* Colonoscopy/CT results.
* Disease event (relapse, metastasis or new primary malignant tumor).
* Survival of subjects.
* Oxaliplatin-induced Peripheral Neuropathy (OXLIPN): Only when oxaliplatin is administered.
* Grade 3-4 adverse drug reactions related to chemotherapy (based on CTCAE v.5.0).
* Serious adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are given explanations about the study objectives and methods, and will express their consent by signing a written agreement to use their personal information.
2. Male and female adult subjects who are ≥ 19 years old.
3. Subjects are confirmed to have primary colon cancer through histological diagnosis and are at *high-risk stage II (T3/4, N0M0) or stage III (any T, N1/2, M0).

   * High-risk stage II is determined when one or more of the following are applicable.

     1. Cancer is at T4 stage (stage IIB,IIC);
     2. Cancer cell differentiation grade is 3 or 4 (poor histologic grade);
     3. Cancer cells are present in lymphatic or blood vessels around the tumor (peritumoral lymphovascular involvement);
     4. Ileus was present during surgery (bowel obstruction at presentation);
     5. Cancer is at T3 stage with localized perforation or there are indeterminate cancer cells residual on the incisal surface. (T3 lesions with localized perforation or close, indeterminate, or positive margins); or,
     6. Cancer cells invaded into the area around the ganglion (perineural invasion).
4. Subjects are decided to require adjuvant chemotherapy including oxaliplatin and/or capecitabine after curative resection (E.g.: FOLFOX, CapeOx or Capecitabine and modified therapies).
5. Subjects' performance status score (ECOG PS) is 2 or lower (0, 1, 2).

Exclusion Criteria:

1. Subjects are diagnosed with other primary cancers that can influence the treatment or prognosis of primary rectal and colon cancers.
2. Subjects are diagnosed with relapsed or secondary colon cancer.
3. Subjects with Stage 0/1 (Tis/1/2, N0M0) or Stage IV (any T, any N, M1) colon cancer.
4. Subjects who are currently on adjuvant chemotherapy after curative resection.
5. Subjects who are receiving palliative chemotherapy.
6. Pregnant and breast-feeding subjects.
7. Subjects who are currently participating in other clinical trials (clinical trials for drugs or medical devices) or are planning to participate in other clinical trials during the duration of this study. However, subjects participating in a noninterventional observational study or a registry study can participate in this study.
8. Other subjects who are not suitable for study participation upon the investigator's decision.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk stage II or stage III primary colon cancer who have received curative resection. Approximately 2,000 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 2013 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Type of adjuvant chemotherapy | through adjuvant chemotherapies completion, an average of 24 weeks
  Type of adjuvant chemotherapy that were used.
Frequency of adjuvant chemotherapy | through adjuvant chemotherapies completion, an average of 12 cycle(FOLFOX: each cycle is 14 days, XELOX or Capacitabine: each cycle is 21 days)
  Frequency of adjuvant chemotherapy that were used.
Disease Free Survival (DFS) | From date of resection surgery until the date of first documented progression, assessed up to 36 months
  Time from the date of resection surgery to the date of first relapse,
Overall Survival (OS) | From date of resection surgery until the date of death, assessed up to 36 months
  Time from the date of resection surgery to the date of death.

SECONDARY OUTCOMES:
Characteristics of relapsed and metastasis cancers and new primary malignant tumor list. | up to 36 months
  Whether locally relapsed, whether metastasis is present, location of metastasis, etc.
Quality of Life Assessment (FACT-C) | Baseline, Month 3 (13 weeks ± 2 weeks), Month 6 (26 weeks ± 2 weeks), Month 12 (52 weeks ± 4 weeks), Month 24 (104 weeks ± 8 weeks), Month 36 (156 weeks ± 8 weeks)
  Subjects will be asked to complete questionnaires to evaluate their quality of life
Quality of Life Assessment (FACT/GOG-NTX-12) | Baseline, Month 3 (13 weeks ± 2 weeks), Month 6 (26 weeks ± 2 weeks), Month 12 (52 weeks ± 4 weeks), Month 24 (104 weeks ± 8 weeks), Month 36 (156 weeks ± 8 weeks)
  Subjects will be asked to complete questionnaires to evaluate their quality of life

OTHER OUTCOMES:
Adverse drug reactions/serious adverse drug reactions | From the date of adjuvant chemotherapy started until the end of follow-up(36 month)
  Overall incidence of grade 3-4 adverse drug reactions/serious adverse drug reactions
Oxaliplatin Induced Peripheral Neuropathy, OXLIPN | From the date of adjuvant chemotherapy started until the end of follow-up(36 month)
  Overall incidence of Oxaliplatin Induced Peripheral Neuropathy, OXLIPN
Performance Status (ECOG) evaluation results | Baseline, Each cycle(FOLFOX: each cycle is 14 days, XELOX or Capacitabine: each cycle is 21 days), Month 3 (13 weeks ± 2 weeks), Month 6 (26 weeks ± 2 weeks), Month 12 (52 weeks ± 4 weeks), Month 24 (104 weeks ± 8 weeks), Month 36 (156 weeks ± 8 weeks)
  Frequency and ratio of ECOG evaluation results will be presented by time point.
Results on weight | Baseline, Each cycle(FOLFOX: each cycle is 14 days, XELOX or Capacitabine: each cycle is 21 days), Month 3 (13 weeks ± 2 weeks), Month 6 (26 weeks ± 2 weeks), Month 12 (52 weeks ± 4 weeks), Month 24 (104 weeks ± 8 weeks), Month 36 (156 weeks ± 8 weeks)
  Descriptive statistics will be presented for the results of weight by time point.
Results on body temperature | Baseline, Each cycle(FOLFOX: each cycle is 14 days, XELOX or Capacitabine: each cycle is 21 days), Month 3 (13 weeks ± 2 weeks), Month 6 (26 weeks ± 2 weeks), Month 12 (52 weeks ± 4 weeks), Month 24 (104 weeks ± 8 weeks), Month 36 (156 weeks ± 8 weeks)
  Descriptive statistics will be presented for the results of body temperature by time point.
Results on pulse | Baseline, Each cycle(FOLFOX: each cycle is 14 days, XELOX or Capacitabine: each cycle is 21 days), Month 3 (13 weeks ± 2 weeks), Month 6 (26 weeks ± 2 weeks), Month 12 (52 weeks ± 4 weeks), Month 24 (104 weeks ± 8 weeks), Month 36 (156 weeks ± 8 weeks)
  Descriptive statistics will be presented for the results of pulse by time point.
Results on blood pressure | Baseline, Each cycle(FOLFOX: each cycle is 14 days, XELOX or Capacitabine: each cycle is 21 days), Month 3 (13 weeks ± 2 weeks), Month 6 (26 weeks ± 2 weeks), Month 12 (52 weeks ± 4 weeks), Month 24 (104 weeks ± 8 weeks), Month 36 (156 weeks ± 8 weeks)
  Descriptive statistics will be presented for the results of blood pressure by time point.

CONTACTS AND LOCATIONS:
Overall Officials: Myung Sook Hong, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea